CLINICAL TRIAL: NCT02694055
Title: Proactive Community Case Management and Child Survival: A Cluster-Randomized Controlled Trial
Brief Title: Trial of Proactive Community Case Management to Reduce Child Mortality
Acronym: Pro-CCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Muso, Inc. (Unknown); Malaria Research and Training Center, Bamako, Mali (Other); University of California, Berkeley (Other); University of Michigan (Other); Instituto Nacional de Salud Publica, Mexico (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Ministère de la Santé et l'Hygiène Publique, Mali (Unknown); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro-CCM-028
Record Dates: First submitted 2016-01-13; First posted 2016-02-29 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Under-five Child Mortality; Access to Health Care
Keywords: Community Health Workers; Community Case Management; Proactive Case Detection; Under-five Child Mortality; Access to Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proactive Community Case Management (ProCCM) (Experimental): Villages assigned to the experimental arm will receive the following health system strengthening interventions: training of primary health centre staff, infrastructure improvements at primary health centre, removal of point-of-care user fees, and the presence of Community Health Workers providing proactive case detection in addition to integrated Community Case Management (ProCCM).
  Interventions: Other: Proactive Community Case Management; Other: Removal of point-of-care user fees; Other: Infrastructure improvements at primary health centre; Other: Training of primary health centre staff
- integrated Community Case Management (iCCM) (Active Comparator): Villages assigned to the active comparator arm will receive the following health system strengthening interventions: training of primary health centre staff, infrastructure improvements at primary health centre, removal of point-of-care user fees, and the presence of Community Health Workers providing passive integrated Community Case Management (iCCM) exclusively at a fixed health post to patients who initiate their own care-seeking.
  Interventions: Other: Integrated Community Case Management; Other: Removal of point-of-care user fees; Other: Infrastructure improvements at primary health centre; Other: Training of primary health centre staff

INTERVENTIONS:
Other: Proactive Community Case Management — CHWs will be trained and deployed to conduct daily active case finding home visits door-to-door for at least two hours each day, with the goal of visiting each household at least two times each month. At these active case finding home visits, CHWs will screen each household of sick children and will offer home pregnancy testing and family planning services to reproductive aged women. For patients they identify, they will offer counselling, diagnostic services, care, accompaniment, and referral according to an iCCM service delivery package.
  Other Names: ProCCM
  Arms: Proactive Community Case Management (ProCCM)
Other: Integrated Community Case Management — CHWs will be trained offer counselling, diagnostic services, care, accompaniment, and referral according to an iCCM service delivery package to patients that visit them at their work post.
  Other Names: iCCM
  Arms: integrated Community Case Management (iCCM)
Other: Removal of point-of-care user fees — User fees will be removed across the catchment areas for both study and control villages. No fees will be charged for care by CHWs or at all primary care centres.
  Other Names: Removal of user fees
Other: Infrastructure improvements at primary health centre — Targeted infrastructure improvements to rehabilitate, expand and equip the capacity of the seven government primary care centres in the study area. Each health center will be equipped with solar power.
  Other Names: Improvements to health centre infrastructure
Other: Training of primary health centre staff — Health center staff will receive targeted training in
  * Integrated management of childhood illness
  * Diagnosis and treatment of simple and severe cases of malaria
  * Helping babies breathe
  * Managing post-partum haemorrhage
  * Gestational dating using frontal height, last menstrual period and ultrasound
  * Family planning counselling and administration of long-acting contraceptives
  * Pharmacy stock management
  * Health center management
  Other Names: Clinical staff training at primary health centres

SUMMARY:
The purpose of this study is to evaluate whether the addition of Proactive Case Detection to Community Case Management will provide an increase in early access to health care and a reduction in deaths among children aged 0-59 months. Integrated Community Case Management is the package of community-based services for children delivered by Community Health Workers (CHW), including diagnosis and treatment of malaria, pneumonia, diarrheal disease and malnutrition. In many iCCM interventions, CHWs are stationed in their villages and available in a passive, reactive manner to provide care to patients who seek them out. This study seeks to determine whether the addition of proactive case detection by CHWs to a standard iCCM intervention (ProCCM), in which they conduct daily door-to-door home visits to find and care for patients, will improve early access to care and reduce child mortality.

Village-clusters will be randomised to receive Integrated Community Case Management (iCCM) from a passive CHW or Proactive Community Case Management (ProCCM) from a CHW that conducts daily active case finding home visits. All villages in both study arms will receive additional interventions that could significantly reduce under-five mortality, including removal of point-of-care fees, clinical staff training at primary health centres, and improvement in primary health centre infrastructure.

All women of reproductive age eligible for inclusion in the study will be surveyed at baseline, and again at 12, 24 and 36 months. The study hypothesis is a significant reduction in child mortality in both study arms, with a significantly larger reduction where there is proactive case detection, or ProCCM, by CHWs. A survey of all women enrolled in the three-year study (eligible and consenting) has 82% power to detect an absolute difference in under-five mortality of 0.75% (a relative difference of 25%) between the two study arms.

DETAILED DESCRIPTION:
The trial is an un-blinded, cluster-randomised controlled trial, with 69 clusters in the intervention arm and 68 clusters in the comparison arm. The cluster is defined as a geographical grouping of homes greater than one kilometre from the next nearest geographical grouping of homes (determined by the cardinal distances between GPS coordinates collected at the public gathering space). In practice, this means a cluster can consist of one village or one hamlet, or a collection of neighbouring villages and/or hamlets.

Clusters were randomised to receive either iCCM from a stationary CHW based at a community health post (control) or ProCCM from a CHW who conducts daily active case-finding home visits for at least two hours a day, six days per week. Randomisation was stratified by distance to PHC (1.0-5.0 km vs. greater than 5.0 km); an additional stratum was defined for all villages where the PHC was located to ensure balanced assignment of PHC villages across arms. Within each strata, villages were randomly assigned to the control or treatment arm using a computer-generated random number, then rank ordered based on this number.

All clusters receive PHC infrastructure improvements and staff training, the removal of user fees at all levels of care, and CHW(s) who provide iCCM of common childhood illnesses in accordance with national and international standards, as well as other community-based services, including a reproductive health package for women of child-bearing age. CHW coverage is based on Mali's national iCCM strategy, which assigns each CHW to an average population of 700 in the southern region. Clusters with less than 200 people and within three kilometres of another cluster assigned to the same study arm share a CHW, provided there is no geographic barrier (i.e. river) between the two clusters and no linguistic barrier for the CHW. CHWs in both arms are required to be on call, available to receive and care for patients who seek them out, 24 hours per day, seven days per week.

The primary outcome is a cluster-level outcome, the under-five mortality rate. It is measured within each cluster as the number of deaths among children under five years of age per 1,000 person-years at risk of mortality. After 36 months, we hypothesize that there will be an absolute difference of 0.75% (or a relative difference of 25%) in under-five child mortality between the two study arms, as measured by the number of deaths per 1,000 person-years among children aged 0 to 59 months. Secondary endpoints include a number of reproductive, maternal, and child health outcomes, as well as access and service delivery outcomes. Secondary objectives also include an economic evaluation of the cost-effectiveness, equity, and affordability at scale of ProCCM compared to iCCM.

An exhaustive census will be administered to the population of the study area (both arms) at baseline. The census will assign a unique identification number to each person surveyed. At each household, a screening will take place to identify women eligible for inclusion. Eligible women identified in the study area will be asked to give written informed consent for their inclusion in the study (or their legal guardians in the case of unemancipated minors). The baseline survey will be administered after consent is obtained. Using the unique census ID number, the same participants will be identified and surveyed again at 12, 24 and 36 months.

The survey tool is excerpted and adapted from Mali's Demographic and Health Survey. The survey tool will collect qualitative and quantitative data on health seeking behaviour and health outcomes. It will include a life-table tracking all live births occurring in the 59 months prior to enrolment and during the 36 months of study follow up. Surveyors will not be members of the villages they survey, nor will they be members of the intervention health care delivery staff. All surveyors will be female, as the survey tool contains potentially sensitive questions on family planning.

Community Health Workers will collect data on the number of active case finding visits they conduct, the number of patients they treat, the delay from symptom onset to treatment onset for each patient, the gestational age at pregnancy diagnosis and first prenatal consultation, and the care services they provide. This data is collected during patient care by CHWs on smartphones using the Medic Mobile for CHWs platform customized for ProCCM. Primary care health centre providers will collect patient care data per village on an electronic medical records system.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age women (aged 15-49 years)
* Permanently living in the study area
* No plans to leave the study area in the subsequent three years
* Written informed consent is obtained

Exclusion Criteria:

* Non-permanent community members (i.e. seasonal migrants)
* Plans to leave study area in the subsequent three years

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 135149 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Difference in the under-five child mortality rate between the two study arms | 36 months
  To assess the effectiveness of ProCCM compared to a passive iCCM intervention, we will compare the three-year under-five mortality rate in treatment versus control clusters collected prospectively in the 12-, 24- and 36-month follow-up surveys.
  We will calculate under-five mortality rate as the number of deaths among children under five years of age per 1,000 person-years of exposure to the risk of mortality for each cluster over the 36-month trial period.

SECONDARY OUTCOMES:
Difference in the infant mortality rate between the two study arms | 36 months
  Infant mortality rate (IMR) is the number of deaths per 1,000 live births among infants aged 0-11 months. We will calculate the IMR over the 36-month trial period.
Difference in the newborn mortality rate between the two study arms | 36 months
  Newborn mortality rate (NMR) is the number of deaths per 1,000 live births among newborns aged 0-28 days. We will calculate the NMR over the 36-month trial period.
Difference in the maternal mortality rate between the two study arms | 36 months
  Maternal mortality ratio (MMR) is the number of deaths among women while pregnant or within 42 days of delivery or termination per 100,000 live births. We calculate the MMR over the 36-month trial period.
Difference in the percentage of women receiving 3 or more doses of SP during their last pregnancy between the two study arms | 36 months
  We will calculate the percentage of women receiving 3 or more doses of Sulfadoxine-Pyrimethamine (SP) during their last pregnancy in the context of Intermittent Preventive Treatment (IPTp) over the 36-month trial period.
Difference in the percentage of under-five children with fever in the prior two weeks who receive testing and/or effective treatment for malaria within 24 hours of symptom onset between the two study arms | 36 months
  The percentage of under-five children with fever in the prior two weeks who receive testing and/or effective treatment for malaria within 24 hours of symptom onset: Among all children who report fever within the two weeks prior to the endline survey (36 months), proportion who report receipt of a malaria rapid diagnostic test (mRDT) and, if the mRDT positive, artemisinin-based combination therapy (arthemeter-lumefantrine) over the 36-month trial period.
Difference in the percentage of children under five with diarrhea in the past two weeks who received zinc and oral rehydration therapy within 24 hours of symptom onset between the two study arms | 36 months
  We will calculate percentage of children under five with diarrhoea in the past two weeks who received zinc and oral rehydration therapy within 24 hours of symptom onset over the 36-month trial period.
Difference in the percentage of children with acute respiratory illness evaluated by a qualified provider within 24 hours of symptom onset between the two study arms | 36 months
  We will calculate the percentage of children with acute respiratory illness (ARI) evaluated by a qualified provider within 24 hours of symptom onset. Among all children who report ARI within the two weeks prior to the endline survey (36 months), proportion who attended a skilled provider within 24 hours of onset of ARI. Skilled providers include CHWs, doctors, nurses, or other providers based at the health center care.
Difference in the percentage of the population accessing CHW or health centre care per month between the two study arms | 36 months
  We will calculate the percentage of the population accessing CHW or health centre care per month over the 36-month trial period.
Difference in the percentage of the population visiting the health centre per month between the two study arms | 36 months
  We will calculate the percentage of the population visiting the health centre per month over the 36-month trial period.
Difference in the percentage of population receiving CHW health care per month between the two study arms | 36 months
  We will calculate the percentage of population receiving CHW health care per month over the 36-month trial period.
Difference in the percentage of the health care seeking population who receive CHW care per month between the two study arms | 36 months
  We will calculate the percentage of the health care seeking population who receive CHW care per month over the 36-month trial period.
Difference in the number of curative consultations per year at the community and health centre level between the two study arms | 36 months
  We will calculate the number of curative consultations per year at the community and health centre level over the 36-month trial period.
Difference in the percentage pregnant women completing four or more prenatal consultations between the two study arms | 36 months
  We will calculate the pregnant women completing four or more prenatal consultations over the 36-month trial period.
Difference in the average gestational age at first prenatal consultation between the two study arms | 36 months
  We will calculate the average gestational age at first prenatal consultation over the 36-month trial period. Alternatively, we will consider percentage of pregnant women with first prenatal consultation in the first trimester over the 36-month trial period.
Difference in the percentage of participants using modern method of a family planning between the two study arms | 36 months
  We will calculate the percentage of participants using a modern method of family planning over the 36-month trial period.

OTHER OUTCOMES:
Cost-effectiveness ratios of i-CCM and Pro-CCM | 36 months
  Cost effectiveness ratios will be presented from three perspectives (i) intervention costs alone, (ii) potential costs/savings to health providers (MoH), (iii) potential societal costs/savings, which includes both health providers and households. Costs to the health care providers and households associated with Pro-CCM and i-CCM will be collected as part of routine trial data collection where possible, with supplementary cost and resource use data collected when necessary. In addition, the economic costs to the health system will be based on detailed cost data from Community Health Workers and health facilities. A standardised costing template will be used in all the sites to record resource use associated with personnel, materials and supplies, equipment, transport, utilities and buildings. Effects will be based on trial outcomes. Specifically, economic evaluation will explore cost of Pro-CCM per disability-adjusted life year saved among children aged 0-59 months.
Equity implications of i-CCM and Pro-CCM | 36 months
  Data on the socio-economic characteristics of study participants will be collected as part of the survey tool, and will include questions that make up the DHS Wealth Index for Mali in order to measure household poverty/wealth. The percentage of children receiving treatment within 24 hours of symptom onset and the survival rate of children 0-59 months will be analysed stratified across wealth quintiles in each trial arm.
Affordability of Pro-CCM at scale | 36 months
  Whether a Pro-CCM program would be affordable to the Ministry of Health will be explored. A simple model forecasting the costs of introducing and sustaining Pro-CCM will be developed and this will run using various 'delivery' (supply) and 'uptake' (demand) scenarios. This model will help to inform decision makers about the affordability of implementing Pro-CCM in their setting.

CONTACTS AND LOCATIONS:
Overall Officials: Ari D Johnson, MD, Study Chair — University California San Francisco; Kassoum Kayantao, PhD, Principal Investigator — Malaria Research & Training Centre, University of Bamako; Nancy S Padian, PhD, Principal Investigator — School of Public Health University of California San Francisco

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available with publication and dissemination of final results after termination of the study in September 2018. However, all IPD made available will be anonymous. IPD includes anonymous quantitative and qualitative data on health seeking behaviour and health outcomes of the study participants.

REFERENCES:
- [Background] Johnson AD, Thomson DR, Atwood S, Alley I, Beckerman JL, Kone I, Diakite D, Diallo H, Traore B, Traore K, Farmer PE, Murray M, Mukherjee J. Assessing early access to care and child survival during a health system strengthening intervention in Mali: a repeated cross sectional survey. PLoS One. 2013 Dec 11;8(12):e81304. doi: 10.1371/journal.pone.0081304. eCollection 2013. PMID 24349053
- [Derived] Ogbuoji O, Shahid M, Zimmerman A, Liu JX, Kayentao K, Whidden C, Treleaven E, Traore C, Sogoba M, Doumbia S, Boettiger DC, Cisse AB, Keita Y, Berthe M, Johnson A. Cost-effectiveness analysis of proactive home visits compared with site-based community health worker care on antenatal care outcomes in Mali: a cluster-randomised trial. BMJ Glob Health. 2024 Dec 27;9(12):e014940. doi: 10.1136/bmjgh-2023-014940. PMID 39732474
- [Derived] Ghosh R, Konipo AN, Treleaven E, Rozenshteyn S, Beckerman J, Whidden C, Johnson A, Kayentao K, Liu J. Factors influencing pregnancy care and institutional delivery in rural Mali: a secondary baseline analysis of a cluster-randomised trial. BMJ Open. 2024 Apr 9;14(4):e084315. doi: 10.1136/bmjopen-2024-084315. PMID 38594181
- [Derived] Whidden C, Kayentao K, Kone N, Liu J, Traore MB, Diakite D, Coumare M, Berthe M, Guindo M, Greenwood B, Chandramohan D, Leyrat C, Treleaven E, Johnson A. Effects of proactive vs fixed community health care delivery on child health and access to care: a cluster randomised trial secondary endpoint analysis. J Glob Health. 2023 Apr 21;13:04047. doi: 10.7189/jogh.13.04047. PMID 37083317
- [Derived] Kayentao K, Ghosh R, Guindo L, Whidden C, Treleaven E, Chiu C, Lassala D, Traore MB, Beckerman J, Diakite D, Tembely A, Idriss BM, Berthe M, Liu JX, Johnson A. Effect of community health worker home visits on antenatal care and institutional delivery: an analysis of secondary outcomes from a cluster randomised trial in Mali. BMJ Glob Health. 2023 Mar;8(3):e011071. doi: 10.1136/bmjgh-2022-011071. PMID 36948531
- [Derived] Oliphant NP, Manda S, Daniels K, Odendaal WA, Besada D, Kinney M, White Johansson E, Doherty T. Integrated community case management of childhood illness in low- and middle-income countries. Cochrane Database Syst Rev. 2021 Feb 10;2(2):CD012882. doi: 10.1002/14651858.CD012882.pub2. PMID 33565123
- [Derived] Whidden C, Treleaven E, Liu J, Padian N, Poudiougou B, Bautista-Arredondo S, Fay MP, Samake S, Cisse AB, Diakite D, Keita Y, Johnson AD, Kayentao K. Proactive community case management and child survival: protocol for a cluster randomised controlled trial. BMJ Open. 2019 Aug 26;9(8):e027487. doi: 10.1136/bmjopen-2018-027487. PMID 31455700
- See also: Muso is an international non-governmental organization working to strengthen the health care system in Mali — http://musohealth.org